CLINICAL TRIAL: NCT00706212
Title: A Comparative Study to Examine the Accuracy of CHOLINE PET CT in the Diagnosis
Brief Title: The Accuracy of CHOLINE PET CT in the Diagnosis of Urological Malignancies
Acronym: GS-PET-2008
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr. Golan Shay, Rabin Medical Center, Urology department
Other Study IDs: GS-PET-2008
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-05

CONDITIONS: Urological Malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
PET CT is one of the imaging tools that are used for staging of urological malignancies.

C11 Choline is a novel isotope with the advantage of its minimal secretion in the urine. This advantage makes it a potentially better metabolic marker then others such as FDG. Preliminary studies showed ~95% sensitivity in the diagnosis of TCC. Our Goal is to continue the evaluation of this method as a diagnostic and follow up tool in different urological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients older then 18 years of age
* Full consciousness and awareness
* suspected to suffer from urological malignancy and a candidate for a surgical procedur

Exclusion Criteria:

* known secondary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rabin Medical center Urological oncology patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-06

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Beilinson hospital, Petah Tikva, Israel